CLINICAL TRIAL: NCT06805084
Title: Trascritti Con Ritenzione Di Sequenze SnoRNA H/ACA Box Come Biomarcatori Per L'estrogeno-dipendenza Nei Carcinomi Della Mammella Luminali B
Brief Title: Transcripts with Retained H/ACA Box SnoRNA Sequences As Biomarkers for Estrogen Dependence in Lum-B Breast Carcinomas
Acronym: H/ACA-ER
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: H/ACA-ER; RC-2024-2790680 (Other Grant/Funding Number: Italian Ministry oh Health)
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-12

CONDITIONS: Breast Adenocarcinoma; Luminal B Breast Cancer
Keywords: oncotype; biomarkers; non coding RNAs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — frozen and formalin fixed tumor specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
RATIONALE:

The primary treatment for estrogen receptor-positive breast cancer relies on estrogen receptor inhibitors. However, responses to hormonal therapy can vary significantly, especially in luminal B breast cancer, necessitating adjuvant chemotherapy for some patients. The Oncotype DX Breast Recurrence Score is the preferred test for determining the most suitable therapy for these patients, providing a Recurrence Score that characterizes the tumor and guides treatment recommendations. Despite its validation, its optimal use in intermediate-risk patients is still unclear.

OBJECTIVES:

Primary Objective:

- Measure whether the expression of mRNAs extracted from paraffin-embedded tissue is associated with the results of the Oncotype DX test.

The primary objective is to evaluate the association between selected mRNA expressions from paraffin-embedded luminal B breast cancer tissue and Oncotype DX test results. This aims to improve current molecular clinical tests and identify new biomarkers for response to anti-estrogen therapy, particularly in luminal B patients with inadequate responses.

Secondary Objectives:

* Assess concordance of mRNA analysis results from paraffin-embedded versus "fresh frozen" tissue.
* Evaluate if mRNA expression levels from paraffin-embedded tissue provide additional characterization for low-risk luminal B patients who do not respond effectively to anti-estrogen therapy.

ENDPOINTS:

Primary Endpoint: Measure potential mRNA biomarker expression values in therapy response groups identified by the Oncotype DX score (low-risk and high-risk).

Secondary Endpoints:

* Measure abundance values of potential mRNA biomarkers from both analysis techniques.
* Calculate treatment response parameters at 36-60 months (Relapse-Free Survival - RFS, Distant Recurrence-Free Survival - DRFS).

STUDY DESIGN:

This study will analyze specific mRNAs in luminal B breast cancer patients by collecting and examining both "fresh frozen" and paraffin-embedded tumor tissues. qPCR will evaluate mRNA expressions of WIPI1, STAT5B, SMAP2, MED24, NCOA3, NCOA7, CCAR1, along with isoforms of EIF4A1, EIF4A2, TAF1D, and UBAP2L. Results will be correlated with Oncotype DX outcomes and diagnostic parameters regarding treatment response. Samples will be collected per standard procedures, ensuring patient treatment aligns with clinical practices, with follow-up data monitored accordingly.

DETAILED DESCRIPTION:
Background and Rationale of the Study The primary approach to treating early-stage estrogen receptor-positive breast cancer involves the use of antitumor drugs (e.g., Tamoxifen) that selectively inhibit estrogen receptors, thereby reducing the risk of recurrence and cancer-related mortality. However, individual responses to hormonal therapy can be highly variable, particularly in luminal B breast cancer, necessitating adjuvant chemotherapy for some patients despite its associated toxic effects. The standard approach to determining the most appropriate therapy for these patients relies on clinical-pathological tumor factors, which, however, have suboptimal prognostic and predictive utility for determining chemotherapy benefits.

To overcome this limitation, several multigene tests have been developed to better stratify prognosis and treatment response. Currently, the standard test for estrogen receptor-positive breast cancer is the Oncotype DX Breast Recurrence Score. This test is based on analyzing the expression of a selected list of genes using RNA extracted from paraffin-embedded patient tumor tissue. It provides a Recurrence Score that characterizes the tumor and guides the recommended therapy. Since 2021, it has been part of the standard of care for luminal B breast cancer patients in Italy. However, its optimal use in intermediate-risk patients remains undefined.

In a recently published study, we identified a specific group of transcripts associated with estrogen response in mammary gland tumors. These transcripts are specific mRNA isoforms that exhibit a unique feature: introns containing the H/ACA box snoRNA (small-nucleolar RNA) sequence. For this reason, we named them snoRT (snoRNA Retain Transcripts). The expression of these transcripts is not only associated with hormone receptor status (both estrogen and progesterone receptors) but is also significantly linked to the survival of hormone receptor-positive patients. Furthermore, we showed that the snoRTs identified in the study interact with other protein-coding transcripts involved in mediating the hormone receptor response. The expression of these transcripts is associated with the survival of breast cancer patients, particularly those with luminal B tumors, making them strong candidates for identifying a potential "molecular signature" associated with luminal B breast cancer outcomes.

Importance of the Study and its Clinical Relevance The recent discoveries mentioned in the background reveal an unexplored role of snoRTs and their interacting protein-coding mRNAs in influencing the dependency of specific tumors on nuclear hormone receptors. Our findings suggest that deregulation of these functions may allow luminal B tumors to escape hormonal dependency, becoming more aggressive and potentially unresponsive to anti-estrogen therapy.

Since estrogen-dependent luminal B tumors sometimes develop characteristics enabling them to overcome hormonal dependency, making them resistant to anti-estrogen therapy, studying this new "molecular signature" and these novel cytoplasmic transcripts appears promising. We propose comparing them with the Oncotype DX test to evaluate whether studying these RNAs can add useful insights for identifying patients unlikely to respond well to anti-estrogen treatments (e.g., those classified as intermediate-risk by the Oncotype DX score). If validated, these new biomarkers could lead to the improvement and refinement of current clinical molecular tests.

The proposed study would represent a significant innovation in the field of biomarkers, as the role of this new class of RNAs (snoRTs) has never been thoroughly investigated and is entirely overlooked by traditional RNA-seq analyses based on genes (due to molecular characteristics related to their localization, transcription, and the maturation of snoRNA genes). The role of snoRTs in regulating gene expression and human diseases remains an unexplored field, and their diagnostic and predictive significance has not been previously considered.

WHAT IS ALREADY KNOWN ABOUT THE TOPIC The primary approach to treating estrogen receptor-positive breast cancer involves using estrogen receptor inhibitors. However, individual responses to hormonal therapy can be highly variable, particularly in luminal B breast cancer, necessitating adjuvant chemotherapy for some patients. To determine the most appropriate therapy for these patients, the preferred test for estrogen receptor-positive breast cancer is the Oncotype DX Breast Recurrence Score. This test provides a Recurrence Score that characterizes the tumor and guides treatment recommendations. Although validated, its optimal use in intermediate-risk patients remains undefined.

WHAT THE STUDY COULD ADD This project aims to define innovative approaches for more precise profiling of luminal B patients who may have developed mechanisms of hormonal independence that often escape detection by conventional tests. Thus, the results of this study could contribute to identifying patients who do not respond to estrogen receptor-targeted therapies. This would enable patients to benefit from more appropriate, and therefore more aggressive, treatment, similar to that offered to high-recurrence-risk patients identified by the Oncotype DX test.

ELIGIBILITY:
Inclusion Criteria:

* Patients with luminal B breast cancer who have undergone the Oncotype DX test at our pathology center, with tissue material available or expected to become available during the enrollment period.
* Age ≥ 18 years
* Informed consent

Exclusion Criteria:

none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be adult female patients with breast cancer who have not previously undergone neoadjuvant chemotherapy and/or hormone therapy and are candidates for surgical removal of breast cancer as part of their standard care pathway. Participants will be selected/enrolled if tissue samples are available or will be obtained within the period between 2019 and 2026.
  The unit responsible for enrollment will be the Oncology Department - Zamagni IRCCS, Azienda Ospedaliero-Universitaria di Bologna Policlinico S. Orsola. Patients will be contacted during a follow-up visit or, if not possible, through an invitation sent by email.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Measure whether the expression of mRNAs extracted from paraffin-embedded tissue is associated with the results of the Oncotype DX test. | 3 years
  The primary objective is to evaluate whether the expression of selected mRNAs extracted from paraffin-embedded luminal B breast cancer tissue is associated with the results of the Oncotype DX test. This comparison aims to refine and improve current molecular clinical tests by assessing their potential as new biomarkers in defining the response to anti-estrogen therapy. This research seeks to identify expression patterns of these RNAs in luminal B patients who exhibit an inadequate response to anti-cancer treatments targeting estrogen receptors.

SECONDARY OUTCOMES:
concordance between fresh and archival material | 1 year
  To verify the concordance of results obtained from the analysis of mRNA extracted from paraffin-embedded tissue with those from frozen tissue, in order to validate and optimize the analysis method.
association with treatment response | 7 years
  To evaluate, in terms of therapy response, whether the analysis of mRNA expression levels extracted from paraffin-embedded tissue in patients who underwent the Oncotype DX test can provide additional characterization of luminal B patients classified as low-risk by the Oncotype DX test but who did not respond effectively to anti-estrogen therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Montanaro, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero Unversitaria di Bologna, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No